CLINICAL TRIAL: NCT03007173
Title: Umbilical Pilonidal Sinus: an Underestimated and Little-known Clinical Entity - Report of Two Cases
Brief Title: Umbilical Pilonidal Sinus: a Case Report
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Principal Investigator, Medical Park Gaziantep Hospital
Other Study IDs: MK-013-UPS
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Umbilical Cyst; Pilonidal Sinus
Keywords: umbilical pilonidal sinus
MeSH Terms: conditions — Urachal Cyst; Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — soft tissue composed of umbilical cyst
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: umbilicus preserving surgery — excision of umbilical complex
  Other Names: pilonidal sinus excision

SUMMARY:
Umbilical pilonidal sinus (UPS) is a rare disease of young, hirsute, dark men with deep navels and poor personal hygiene; however, it can be seen in females. UPS could easily be misdiagnosed and mistreated due to its rarity and lack of awareness in physicians. Diagnosis is easy to establish with physical examination and a detailed history. Treatment is generally depending on the severity of the disease, ranging from good personal hygiene to surgical excision of umbilical complex. The treatment of choice for chronic, intermittent cases is surgical removal of the affected portion; paying special attention to cosmetic appearance especially in female patients. In this report, we present two cases of UPS, one in a man and one in a woman with the explanation of its etiopathogenesis and surgical treatment.

DETAILED DESCRIPTION:
Introduction: Umbilical pilonidal sinus (UPS) is a rare disease of young, hirsute, dark men with deep navels and poor personal hygiene. It is being diagnosed and reported more frequently; however, there is still no consensus regarding its best treatment options.

Presentation of cases: In this report, we present two cases of UPS, one in a man and one in a woman who had typical symptoms with pain, swelling and intermittent malodorous discharge from the umbilicus. They had small sinus openings with hair protruding deep in the navel. Because patients had previous history of failed conservative treatments an umbilicus preserving surgery was performed for both cases.

ELIGIBILITY:
Inclusion Criteria:

* no limitation

Exclusion Criteria:

* patients followed-up less than 2 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No limitation for age, gender, ethnicity
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
cure rate | within 2 years of follow-up
  Primary outcome was the cure rate. Absence of recurrence within two year after the first treatment was considered as a cure.
  Recurrence was defined as the appearance of a new, active discharging sinus or granulation tissue with/without a bit of hairs in the deep of the umbilicus within two years after therapy.

SECONDARY OUTCOMES:
healing time | within the postoperative 1 month
  the time form initial treatment to healing the wound and/or sinus and/or granulation tissue and no any sign of drainage with no longer need for dressing and wound care in either treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Principal Investigator — Medical Park Hospital
Locations (1):
- Mehmet Kaplan, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan M, Ozcan O, Kaplan FC, Yalcin HC, Salman B. Conservative vs Surgical Interventions for Umbilical Pilonidal Sinus: A Multicenter, Double-Blind, Prospective, Randomized Clinical Trial. J Am Coll Surg. 2016 May;222(5):878-89. doi: 10.1016/j.jamcollsurg.2016.01.056. Epub 2016 Feb 23. PMID 27016906